CLINICAL TRIAL: NCT03453008
Title: Study of Spastic Cocontractions and Limitation of Active Movements of the Upper Limb Before and After Treatment During Injection of Botulinum Toxin in Patients After Stroke
Brief Title: Spastic Cocontractions and Limitation of Active Movements Before and After Treatment During Injection of Botulinum Toxin
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0191; 2017-A01616-47 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Cerebrovascular Accident; Stroke
Keywords: Cerebrovascular Accident; Botulinum toxin A; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: elbow extension, electromyography — Two evaluations before the toxin injection (T0 and T1), to quantify cocontractions and to determine the toxin injection pattern.
  The first evaluation (T0) will be carried out within a period of between 1 month and 15 days before the injection. This evaluation makes it possible to pose the indication for the realization of injection of Botulinum Toxin A (TBA).
  The second evaluation (T1) will be performed on the day of the injection to specify the muscle targets to be injected.
  The first evaluation is a Clinical evaluation and second is Instrumental evaluation

SUMMARY:
Following a stroke , 55% of the patients do not recover any traction of the upper limb and 30% a residual motricity not allowing a functional grip. For this last group of patients, there are major therapeutic issues to restore a functional grip.

The aim of the study is to relieved the spastic cocontractions before and after usual injection of botulinum toxin A at stroke patient.

DETAILED DESCRIPTION:
Descriptive study of spastic cocontraction index before and after botulinum toxin A injections during active elbow extension in chronic vascular hemiplegic patients.

The spastic cocontraction score will be compared between T1 (before the Botulinum toxin A injection) and T2 (4 weeks after the botulinum toxin A injection in the elbow flexors).

There is no control group. The patient is his own witness: the non-paretic side is considered as the physiological reference in terms of the level of spastic cocontractions.

Botulinum toxin A injections are performed in routine clinical practice in the Physical Medicine and Rehabilitation Department, following the recommendations in force. This treatment has been shown to be effective on spasticity in several high-level studies. The reduction of spasticity, evaluated clinically (Tardieu and Ashworth scale), is a criterion of efficacy of botulinum toxin A injections.

The evaluation of the effectiveness of botulinum toxin A injections on the other components of muscular hyperactivity, such as the reduction of spastic cocontraction during active movements, is poorly performed in clinical and clinical research. This protocol includes specific assessments to evaluate the evolution of spastic cocontraction.

ELIGIBILITY:
Inclusion Criteria:

* Having notified his non-opposition to participate in the search
* Ischemic or hemorrhagic stroke of more than 6 months, cortical and / or subcortical;
* Indication to the realization of an injection of Botulinum Toxin A in the flexor muscles of the elbow according to the usual clinical criteria: presence of a functional complaint or aesthetic expressed by the patient and related to hyperactivity muscular (spasticity or cocontraction) on the flexor muscles elbow, which is a focal treatment by injection of botulinum toxin;
* Possibility of active extension of elbow> 20 °;
* Patients naive to Botulinum Toxin A or more than 4 months of a first injection of Botulinum Toxin A, having targeted the elbow flexors.

Exclusion Criteria:

* Passive limitation of elbow extension> 30 °;
* Pain when performing active movements of flexion / extension of the elbow
* Cognitive impairment limiting the comprehension of three basic instructions (proof test of the 3 papers of the MMS);
* Evolutionary or decompensated neurological pathology; Ischemic or haemorrhagic stroke of less than 6 months;
* General contraindication to the production of botulinum toxin; history of myasthenia gravis, Lambert Eaton syndrome; history of neuromuscular disease; surgery with curarization for less than 1 month; treatment with aminoglycoside, aminoquinoline or cyclosporine
* Legal incapacity (safeguard of justice, guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Ischemic or hemorrhagic stroke of more than 6 months, cortical and / or subcortical and an who can have a Botulinum Toxin A injection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of spastic cocontraction index during active elbow extension | 2 hours
  Measurement of spastic cocontraction index during active elbow extension, obtained from the electromyography signal of the extensor and flexor muscles of the elbow paretic side, between T1 and T2 (before / after the injection of Botulinum Toxin A).

SECONDARY OUTCOMES:
Sensory balance of the upper limb | 2 hours
  The Erasmus Modified Nottingham Assessment (EmNSA), validated in English, allows a comprehensive evaluation of the superficial epicritic, proprioceptive sensitivity and stereognosis of the entire upper limb in the hemiplegic patient.
Evaluation of the voluntary muscular force | 2 hours
  Held and Pierrot-Deseilligny scale, which abstracts from the notions of gravity and range of motion.
Evaluation of spasticity | 2 hours
  It is evaluated by the Tardieu scale. The analysis will consist of studying the evolution of the muscular reaction and its angle of onset (Tardieu scale) during each of the clinical evaluations.
Limitation of Active Motion Angle Elbow Extension | 2 hours
  Limitation of Active Motion Angle (LAMA) is the clinical measure of the consequences of a spastic cocontraction in a patient. To calculate it, we subtract the maximum elbow extension angle obtained during the PASSIVE stretch of the muscles at the maximum elbow extension angle obtained during a voluntary ACTIVE contraction. As part of the protocol, the LAMA will be instrumentally measured with the 3D kinematic system (Optitrack).
  This data is expressed in gross value (in degrees) or in percentage (depending on the maximum amplitude obtained during passive stretching).
Fugl-Meyer score (motor selectivity) | 2 hours
  The Fugl-Meyer Motor Function Assessment (FMA-Motor), based on the motor recovery scheme described by Brunnstrom (1975), is a scale of evaluation of voluntary reference motor function in the cerebral adult, often used in research and development in clinical practice. The FMA-Motor part of the upper limb is rated 66. It has high validity, reliability and sensitivity to change.
Functional abilities with the Wolf Motor Function Test score | 2 hours
  Functional abilities with the Wolf Motor Function Test validated in more than 16 languages (including French) since 2013, is a standardized scale evaluating upper limb capacities in cerebral palsy adults. Originally designed by Steven Wolf (1987) to quantify the effects of stress-induced therapy, this tool is often used in research protocols in the acute and chronic phase brain. The scale consists of performing 17 standardized tests, classified in order of increasing complexity, which solicit the proximal joints

CONTACTS AND LOCATIONS:
Overall Officials: David Gasq, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No